CLINICAL TRIAL: NCT01163292
Title: Humira 40 mg/0.8 mL Syringe for Subcutaneous Injection - Special Investigation (Follow-up Survey of the Study of Adalimumab (D2E7) for Prevention of Joint Destruction in Patients With Rheumatoid Arthritis in Japan (M06-859)]
Brief Title: Special Investigation (Follow-up Survey of the Study of Adalimumab (D2E7) for Prevention of Joint Destruction in Patients With Rheumatoid Arthritis in Japan (M06-859 (NCT00870467))
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-069
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2013-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adalimumab: Participants who continued adalimumab treatment after completion of Study NCT00870467 (M06-859)
- Non-Adalimumab: Participants who discontinued adalimumab treatment after completion of Study NCT00870467(M06-859)

SUMMARY:
The present survey was conducted to evaluate the effectiveness and safety of treatment with adalimumab during the 52-week period following completion of the treatment period in Study NCT00870467 (M06-859) in participants who continued treatment with adalimumab for 52 weeks.

DETAILED DESCRIPTION:
This survey was conducted to assess the risk and benefit of continuing or discontinuing biological therapy with adalimumab (Humira) during the 52-week period following completion of the treatment period in Study NCT00870467 (M06-859).

ELIGIBILITY:
Inclusion Criteria:

* The participants were patients who continued treatment with adalimumab until the end of the treatment period in the NCT00870467(M06-859) study and provided informed consent to participate in the present follow-up survey.

Exclusion Criteria:

* Participants who used biological agents other than adalimumab after the period of treatment in the NCT00870467(M06-859) study were excluded from the present follow-up study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants were patients who continued treatment with adalimumab until the end of the treatment period in the NCT00870467(M06-859) study.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2010-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aki Kuroki, Study Director — AbbVie
Locations (75):
- Japan (75):
  - Site Reference ID/Investigator# 54680, Anjo
  - Site Reference ID/Investigator# 54677, Aomori
  - Site Reference ID/Investigator# 54516, Chiba
  - Site Reference ID/Investigator# 54660, Chiba
  - Site Reference ID/Investigator# 54683, Chiba
  - Site Reference ID/Investigator# 54521, Fukuoka
  - Site Reference ID/Investigator# 39854, Gifu
  - Site Reference ID/Investigator# 54666, Hamamatsu
  - Site Reference ID/Investigator# 54682, Hiroshima
  - Site Reference ID/Investigator# 54669, Hyōgo
  - Site Reference ID/Investigator# 54674, Hyōgo
  - Site Reference ID/Investigator# 54653, Ibaraki
  - Site Reference ID/Investigator# 54670, Kagoshima
  - Site Reference ID/Investigator# 54692, Kagoshima
  - Site Reference ID/Investigator# 54679, Kawagoe
  - Site Reference ID/Investigator# 59580, Kawagoe
  - Site Reference ID/Investigator# 54662, Kawasaki
  - Site Reference ID/Investigator# 54693, Kirishima
  - Site Reference ID/Investigator# 54671, Kitakyushu
  - Site Reference ID/Investigator# 54643, Kumamoto
  - Site Reference ID/Investigator# 59583, Kyoto
  - Site Reference ID/Investigator# 59582, Maebashi
  - Site Reference ID/Investigator# 39849, Matsumoto
  - Site Reference ID/Investigator# 54520, Matsuyama
  - Site Reference ID/Investigator# 54644, Miyazaki
  - Site Reference ID/Investigator# 54645, Morioka
  - Site Reference ID/Investigator# 54654, Nagano
  - Site Reference ID/Investigator# 54656, Nagaoka
  - Site Reference ID/Investigator# 63052, Nagasaki
  - Site Reference ID/Investigator# 54667, Nagoya
  - Site Reference ID/Investigator# 54673, Nagoya
  - Site Reference ID/Investigator# 54649, Nara
  - Site Reference ID/Investigator# 39844, Niigata
  - Site Reference ID/Investigator# 39847, Okayama
  - Site Reference ID/Investigator# 54681, Okayama
  - Site Reference ID/Investigator# 39846, Osaka
  - Site Reference ID/Investigator# 54518, Osaka
  - Site Reference ID/Investigator# 54675, Ōita
  - Site Reference ID/Investigator# 54646, Rifu
  - Site Reference ID/Investigator# 54661, Sagamihara, Kanagawa
  - Site Reference ID/Investigator# 54514, Saitama
  - Site Reference ID/Investigator# 54689, Saitama
  - Site Reference ID/Investigator# 25922, Sapporo
  - Site Reference ID/Investigator# 39850, Sapporo
  - Site Reference ID/Investigator# 54651, Sapporo
  - Site Reference ID/Investigator# 54652, Sapporo
  - Site Reference ID/Investigator# 54522, Sasebo
  - Site Reference ID/Investigator# 54650, Setouchi
  - Site Reference ID/Investigator# 39851, Shimotsuke
  - Site Reference ID/Investigator# 39845, Shizuoka
  - Site Reference ID/Investigator# 54517, Shizuoka
  - Site Reference ID/Investigator# 59579, Takamatsu
  - Site Reference ID/Investigator# 54655, Takasaki
  - Site Reference ID/Investigator# 54519, Tenri
  - Site Reference ID/Investigator# 54515, Tokorozawa
  - Site Reference ID/Investigator# 39842, Tokyo
  - Site Reference ID/Investigator# 39852, Tokyo
  - Site Reference ID/Investigator# 39853, Tokyo
  - Site Reference ID/Investigator# 54647, Tokyo
  - Site Reference ID/Investigator# 54657, Tokyo
  - Site Reference ID/Investigator# 54658, Tokyo
  - Site Reference ID/Investigator# 54678, Tokyo
  - Site Reference ID/Investigator# 54688, Tokyo
  - Site Reference ID/Investigator# 59581, Tokyo
  - Site Reference ID/Investigator# 54672, Tomigusuku
  - Site Reference ID/Investigator# 54648, Toyama
  - Site Reference ID/Investigator# 54691, Toyama
  - Site Reference ID/Investigator# 54690, Toyoake
  - Site Reference ID/Investigator# 54676, Toyohashi
  - Site Reference ID/Investigator# 54668, Tsu
  - Site Reference ID/Investigator# 39843, Yokohama
  - Site Reference ID/Investigator# 54663, Yokohama
  - Site Reference ID/Investigator# 54664, Yokohama
  - Site Reference ID/Investigator# 54665, Yokohama
  - Site Reference ID/Investigator# 54659, Yotsukaidō

REFERENCES:
- [Derived] Tanaka Y, Yamanaka H, Ishiguro N, Miyasaka N, Kawana K, Hiramatsu K, Takeuchi T. Adalimumab discontinuation in patients with early rheumatoid arthritis who were initially treated with methotrexate alone or in combination with adalimumab: 1 year outcomes of the HOPEFUL-2 study. RMD Open. 2016 Feb 18;2(1):e000189. doi: 10.1136/rmdopen-2015-000189. eCollection 2016. PMID 26925252
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab: Participants who continued adalimumab treatment after completion of Study NCT00870467(M06-859)
- Non-Adalimumab: Participants who discontinued adalimumab treatment after completion of Study NCT00870467 (M06-859)
Period: Overall Study
Arm/Group | Adalimumab | Non-Adalimumab
Started | 106 | 114
Completed | 65 | 92
Not Completed | 41 | 22
Not completed — Lack of Efficacy | 9 | 0
Not completed — Adverse Event | 6 | 0
Not completed — Initiation of biological therapy | 0 | 15
Not completed — Sufficient response to adalimumab | 8 | 0
Not completed — Refusal to receive adalimumab | 7 | 0
Not completed — Economic reasons | 6 | 0
Not completed — No further visits | 5 | 7

BASELINE CHARACTERISTICS:
Population: All participants registered
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab | Non-Adalimumab | Total
Number analyzed (Participants) | 106 | 114 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (13.0) | 54.7 (12.3) | 55.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 92 | 179
  Male | 19 | 22 | 41
Body weight [Mean (Standard Deviation); unit: kg] | 55.46 (8.99) | 57.53 (11.08) | 56.53 (10.16)
Rheumatoid arthritis duration [Mean (Standard Deviation); unit: years] | 1.290 (0.428) | 1.316 (0.438) | 1.303 (0.433)
Prior Disease Modifying Anti-Rheumatic Drug (except methotrexate) [Number; unit: participants]
  Yes | 58 | 51 | 109
  No | 48 | 63 | 111
Concomitant Glucocorticoid Use [Number; unit: participants]
  Yes | 33 | 30 | 63
  No | 73 | 84 | 157
Rheumatoid Factor [Number; unit: participants]
  Positive | 60 | 71 | 131
  Negative | 46 | 43 | 89
Health Assessment Questionnaire Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — Participants assessed their ability to perform the following tasks: 1) dress/groom; 2) arise; 3) eat; 4) walk; 5) reach; 6) grip; 7) maintain hygiene; and 8) maintain daily activity. Participants assessed their ability to do these tasks over the past week by marking their response on a questionnaire. Possible responses/scores included the following: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3).
  units on a scale | 0.29 (0.34) | 0.25 (0.33) | 0.27 (0.34)
Disease Activity Score [Mean (Standard Deviation); unit: units on a scale] — The Disease Activity Score (DAS28) is a combined index used to measure disease activity in patients with rheumatoid arthritis. Calculation of the DAS28 score used the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity, and the erythrocyte sedimentation rate (ESR). DAS 28 (ESR) scores range from 0 (no disease activity) to 9 (maximal disease activity).
  units on a scale | 2.89 (1.10) | 2.74 (1.11) | 2.81 (1.11)
Modified Total Sharp Score (mTSS) [Mean (Standard Deviation); unit: units on a scale] — Modified Total Sharp Score (mTSS) is a method of assessing radiographs, used in evaluation of inhibition of joint destruction of disease. Digitized X-rays of hands and feet were obtained, then scored in a blinded manner: for erosion (0 [no damage] to 5 [complete collapse or total destruction of joint]) and for joint space narrowing (0 [no damage] to 4 [complete luxation of joint]). Sum of scores was given as total mTSS (0 [normal] to 380 [maximal disease]).
  units on a scale | 15.61 (22.19) | 16.47 (22.30) | 16.05 (22.20)
Matrix Metalloprotease (MMP-3) [Mean (Standard Deviation); unit: ng/mL] — Matrix metalloprotease level in serum
  ng/mL
    Male | 149.95 (114.81) | 113.70 (135.15) | 130.50 (125.92)
    Female | 86.94 (113.09) | 88.88 (182.09) | 87.94 (152.09)

OUTCOME MEASURES:

1. Primary Outcome: Disease Activity Score (DAS28)
Description: The Disease Activity Score (DAS28) is a combined index used to measure disease activity in participants with rheumatoid arthritis. Calculation of the DAS28 score used the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity, and the erythrocyte sedimentation rate (ESR). DAS 28 (ESR) scores range from 0 (no disease activity) to 9 (maximal disease activity); decrease is indicative of improvement in disease activity.
Time Frame: Weeks 0, 26, and 52
Population: All participants with post-baseline DAS28 data, using last-observation-carried forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab | Non-Adalimumab
Number analyzed (Participants) | 91 | 95
units on a scale
  Week 0 | 2.93 (1.05) | 2.73 (1.04)
  Week 26 | 2.72 (1.12) | 3.17 (1.11)
  Week 52 | 2.70 (1.08) | 3.20 (1.24)
Statistical Analysis 1: Comparison: Adalimumab vs Non-Adalimumab; Week 0; Test type: Superiority or Other; p = 0.144, Wilcoxon Rank Sum
Statistical Analysis 2: Comparison: Adalimumab vs Non-Adalimumab; Week 26; Test type: Superiority or Other; p = 0.004, Wilcoxon Rank Sum
Statistical Analysis 3: Comparison: Adalimumab vs Non-Adalimumab; Week 52; Test type: Superiority or Other; p = 0.006, Wilcoxon Rank Sum

2. Secondary Outcome: Matrix Metalloprotease-3 (MMP-3)
Description: MMP-3 level in serum. Positive = >/= 121.0 ng/mL (male) and 59.7 ng/mL (female)
Time Frame: Weeks 0, 26, and 52
Population: All participants with post-baseline MMP-3 data, using LOCF imputation method
Measure: Number; unit: units on a scale
Arm/Group | Adalimumab | Non-Adalimumab
Number analyzed (Participants) | 93 | 96
units on a scale
  Week 0 Positive | 36 | 30
  Week 0 Negative | 57 | 66
  Week 26 Positive | 34 | 35
  Week 26 Negative | 59 | 61
  Week 52 Positive | 21 | 43
  Week 52 Negative | 72 | 53
Statistical Analysis 1: Comparison: Adalimumab vs Non-Adalimumab; Week 0; Test type: Superiority or Other; p = 0.290, Fisher Exact
Statistical Analysis 2: Comparison: Adalimumab vs Non-Adalimumab; Week 26; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: Adalimumab vs Non-Adalimumab; Week 52; Test type: Superiority or Other; p = 0.001, Fisher Exact

3. Secondary Outcome: Modified Total Sharp Score (mTSS) Change From Week 0 to Week 52
Description: Modified Total Sharp Score (mTSS) is a method of assessing radiographs used in evaluation of inhibition of joint destruction of disease. Digitized X-rays of hands and feet were obtained, then scored in a blinded manner: for erosion (0 [no damage] to 5 [complete collapse or total destruction of joint]) and for joint space narrowing (0 [no damage] to 4 [complete luxation of joint]). Sum of scores was given as total mTSS (0 [normal] to 380 [maximal disease]). Large positive change in mTSS indicates disease progression; small positive/no change indicates slowing/halting of disease progression.
Time Frame: Week 0 to Week 52
Population: All participants with post-baseline mTSS data, using LOCF imputation method
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab | Non-Adalimumab
Number analyzed (Participants) | 86 | 96
units on a scale | 0.8 (3.9) | 0.6 (1.8)
Statistical Analysis 1: Comparison: Adalimumab vs Non-Adalimumab; Test type: Superiority or Other; p = 0.335, Wilcoxon Rank Sum

4. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: Participants assessed their ability to perform the following tasks: 1) dress/groom; 2) arise; 3) eat; 4) walk; 5) reach; 6) grip; 7) maintain hygiene; and 8) maintain daily activity. Participants assessed their ability to do these tasks over the past week by marking their response on a questionnaire. Possible responses/scores included the following: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Negative mean changes from baseline in the disability index of the HAQ-DI indicated improvement.
Time Frame: Weeks 0, 26, and 52
Population: All participants with post-baseline HAQ-DI data, using LOCF imputation method
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab | Non-Adalimumab
Number analyzed (Participants) | 85 | 82
units on a scale
  Week 0 | 0.27 (0.32) | 0.24 (0.33)
  Week 26 | 0.20 (0.32) | 0.24 (0.36)
  Week 52 | 0.20 (0.29) | 0.26 (0.39)
Statistical Analysis 1: Comparison: Adalimumab vs Non-Adalimumab; Week 0; Test type: Superiority or Other; p = 0.266, Wilcoxon Rank Sum
Statistical Analysis 2: Comparison: Adalimumab vs Non-Adalimumab; Week 26; Test type: Superiority or Other; p = 0.440, Wilcoxon Rank Sum
Statistical Analysis 3: Comparison: Adalimumab vs Non-Adalimumab; Week 52; Test type: Superiority or Other; p = 0.609, Wilcoxon Rank Sum

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Adverse events (AEs) were collected from week 0 till the end of the study. Please see Adverse Event section below for more details.
Time Frame: Week 0 to Week 52
Population: All participants registered
Measure: Number; unit: participants
Arm/Group | Adalimumab | Non-Adalimumab
Number analyzed (Participants) | 106 | 114
participants | 51 | 39

ADVERSE EVENTS:
Time Frame: Week 0 to Week 52
Arm/Group | Adalimumab | Non-Adalimumab
Serious Adverse Events (participants affected / at risk) | 5/106 | 3/114
Other Adverse Events (participants affected / at risk) | 46/106 | 36/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=106) | Non-Adalimumab (N=114)
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Scar (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=106) | Non-Adalimumab (N=114)
Cataract (Eye disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 1
Injection site reaction (General disorders) | 4 | 0
Pyrexia (General disorders) | 2 | 0
Liver disorder (enzyme elevation) (Hepatobiliary disorders) | 1 | 2
Bronchitis (Infections and infestations) | 3 | 2
Gastroenteritis (Infections and infestations) | 3 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 13 | 8
Pharyngitis (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 1 | 1
Oral herpes (Infections and infestations) | 2 | 3
Fall (Injury, poisoning and procedural complications) | 2 | 0
White blood cell count decreased (Investigations) | 2 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 3
Headache (Nervous system disorders) | 3 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Hypertension (Vascular disorders) | 1 | 2
Angina pectoris (Cardiac disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Punctate keratitis (Eye disorders) | 0 | 1
Xerophthalmia (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Chelitis (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Pancreatic enlargement (Gastrointestinal disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 1
Driug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 1
Genital candidiasis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Bronchitis bacterial (Infections and infestations) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Breast discomfort (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash generalized (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.